CLINICAL TRIAL: NCT05445778
Title: Randomized, Multicenter, Open-label, Phase 3 Study of Mirvetuximab Soravtansine in Combination With Bevacizumab Versus Bevacizumab Alone as Maintenance Therapy for Patients With FRα-high Recurrent Platinum-sensitive Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancers Who Have Not Progressed After Second Line Platinum-based Chemotherapy Plus Bevacizumab
Brief Title: Mirvetuximab Soravtansine With Bevacizumab Versus Bevacizumab as Maintenance in Platinum-sensitive Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer
Acronym: GLORIOSA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0421; 2022-501606-35 (Other: EU CT)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum-sensitive; Folate-receptor alpha expression; Antibody-drug conjugate; Cancer; Ovarian Neoplasma; Recurrent Platinum-Sensitive; High-Grade Ovarian; ADC; Adult
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — mirvetuximab soravtansine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Mirvetuximab Soravtansine (MIRV) plus Bevacizumab
  Interventions: Drug: Mirvetuximab soravtansine plus Bevacizumab
- Arm 2 (Active Comparator): Bevacizumab monotherapy
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Mirvetuximab soravtansine plus Bevacizumab — Participants will receive MIRV 6.0 mg/kg adjusted ideal body weight (AIBW) plus Bevacizumab 15mg/kg every 3 weeks
  Other Names: MIRV
  Arms: Arm 1
Drug: Bevacizumab — Participants will receive Bevacizumab 15mg/kg every 3 weeks
  Arms: Arm 2

SUMMARY:
GLORIOSA is a Phase 3 multicenter, open label study designed to evaluate the safety and efficacy of mirvetuximab Soravtansine + Bevacizumab as maintenance therapy in participants with platinum-sensitive ovarian, primary peritoneal or fallopian tube cancers with high folate receptor-alpha (FRα) expression.

DETAILED DESCRIPTION:
Mirvetuximab Soravtansine (MIRV) is an investigational antibody drug conjugate designed to selectively kill cancer cells. The antibody (protein) part of MIRV targets tumors by delivering a cell-killing drug to the tumor cells carrying a tumor-associated protein called folate receptor alpha (FRα). It is being developed as maintenance therapy for the treatment of subjects with recurrent platinum-sensitive, highgrade epithelial ovarian, primary peritoneal, or fallopian tube cancers with high folate receptor-alpha expression. Patients must have confirmation of FRα positivity by the Ventana FOLR1 Assay.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women >/=18 years old
2. Confirmed diagnosis of high-grade serous epithelial ovarian, primary peritoneal, or fallopian tube cancer
3. Confirmed high FRα expression by regulatory-agency approved Ventana FOLR1 (FOLR1-2.1)
4. Relapsed disease after frontline (first-line) platinum-based chemotherapy and must be plantinum-sensitive
5. Willing and able to sign the informed consent form (ICF) and adhere to protocol requirements
6. Negative pregnancy test and willing to use highly effective contraceptive method(s) while on study medication and for at least 7 months after the last dose of MIRV and 6 months after the last dose of bevacizumab

Exclusion Criteria:

1. Endometrioid, clear cell, mucinous, or sarconmatous histology; mixed tumors containing any of the above or low grade/borderline ovarian tumor
2. More than one line of prior chemotherapy before current/planned triplet therapy
3. PD (progressive disease) while on or following platinum-based therapy
4. Prior or whole-pelvis or wide-field radiotherapy
5. > Grade 1 peripheral neuropathy
6. History of or concurrent ocular disorders
7. Grade 4 thromboembolic events
8. Not appropriate for bevacizumab treatment
9. Requiring use of folate-containing supplements
10. Prior hypersensitivity to monoclonal antibodies
11. Pregnant or breatfeeding women
12. Received prior MIRV or other FRα-targeting agents
13. Untreated or symptomatic central nervous system metastases
14. History of other malignancy within 3 years prior to signing study consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 520 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Assess Progression-free survival (PFS) | Up to 4 years
  Progression-free survival defined as assessed by BICR per RECIST v1.1, defined as the time from date of randomization until BICR-assessed PD or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Assess Overall survival (OS) | Up to 10 years
  Overall survival (OS), defined as the time from randomization to death
Assess Safety and tolerability | Up to 10 years
  Adverse events (AEs) will be evaluated according to the NCI CTCAE v5
Assess time to second disease progression (PFS2) | Up to 10 years
  Second disease progression (PFS2) defined as the time from date of randomization until second disease progression or death, whichever occurs first
Assess Objective Response Rate (ORR) | Up to 10 years
  Objective response includes best response of complete response (CR) or partial response (PR).
Assess Duration of response (DOR) | Up to 10 years
  DOR as assessed by the investigator and by BICR in patients who have measurable disease per RECIST v1.1 at randomization and achieved a confirmed response of CR or PR after maintenance therapy"
Assess Disease-free survival (DFS) | Up to 10 years
  DOR as assessed by the investigator and by BICR in patients who have no measurable disease per RECIST v1.1 at randomization
CA-125 response | Up to 10 years
  Serum CA-125 response determined using the GCIG criteria
Patient-reported outcome health-related quality of life (HRQoL) of disease-related symptoms using the NCCN-FACT Ovarian Symptom Index (NFOSI-18) DRS-P (disease-related symptom subscale - physical). | Up to 10 years
  A questionnaire assessing the health of patients with ovarian cancer.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (260):
- United States (71):
  - Usa Mitchell Cancer Institute /ID# 269661, Mobile, Alabama
  - Honorhealth Virginia G. Piper Cancer Care Network - Biltmore /ID# 269987, Phoenix, Arizona
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 269573, Irvine, California
  - Moores Cancer Center at UC San Diego /ID# 269564, La Jolla, California
  - University Of California Irvine Medical Center /ID# 269572, Orange, California
  - Stanford Women'S Cancer Center /ID# 269552, Palo Alto, California
  - Kaiser Permanente Zion Medical Center /ID# 269537, San Diego, California
  - Kaiser Permanente - San Diego Medical Center /ID# 269540, San Diego, California
  - Kaiser Permanente - San Marcos Medical Offices /ID# 269542, San Marcos, California
  - Olive View-Ucla Medical Center /ID# 269584, Sylmar, California
  - John Muir Health - Walnut Creek Medical Center /ID# 269575, Walnut Creek, California
  - Broward General Medical Center /ID# 269577, Fort Lauderdale, Florida
  - Regional Cancer Center /ID# 269558, Fort Myers, Florida
  - Baptist Md Anderson Cancer Center - Jacksonville - Palm Avenue /ID# 269560, Jacksonville, Florida
  - Mount Sinai Medical Center /ID# 269582, Miami, Florida
  - Sarasota Memorial Hospital /ID# 269526, Sarasota, Florida
  - Northside Hospital /ID# 269660, Atlanta, Georgia
  - Rush University Medical Center /ID# 269583, Chicago, Illinois
  - University of Chicago Medical Center /ID# 269546, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center /ID# 269110, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital /ID# 269107, Indianapolis, Indiana
  - University of Iowa /ID# 269566, Iowa City, Iowa
  - The University of Kansas Cancer Center - Westwood /ID# 269106, Westwood, Kansas
  - Baptist Health Lexington /ID# 269568, Lexington, Kentucky
  - University of Kentucky Chandler Medical Center /ID# 269536, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - New Orleans /ID# 269559, New Orleans, Louisiana
  - Ochsner Medical Center - Jefferson Highway /ID# 269530, New Orleans, Louisiana
  - Maine Medical Center - Scarborough Campus /ID# 269555, Scarborough, Maine
  - Johns Hopkins Hospital /ID# 269579, Baltimore, Maryland
  - Sinai Hospital Of Baltimore /ID# 269567, Manchester, Maryland
  - GBMC Cancer Center /ID# 269561, Towson, Maryland
  - Tufts Medical Center /ID# 269547, Boston, Massachusetts
  - Baystate Medical Center /ID# 269544, Springfield, Massachusetts
  - Corewell Health /ID# 269562, Grand Rapids, Michigan
  - Minnesota Oncology - Coon Rapids Clinic /ID# 269550, Coon Rapids, Minnesota
  - Nebraska Methodist Hospital /ID# 269580, Omaha, Nebraska
  - The Center Of Hope /ID# 269528, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 269576, Lebanon, New Hampshire
  - John Theurer Cancer Center /ID# 269109, Hackensack, New Jersey
  - The Valley Hospital /ID# 269548, Paramus, New Jersey
  - Holy Name Medical Center /ID# 269543, Teaneck, New Jersey
  - New York Oncology Hematology - Albany Cancer Center /ID# 269565, Albany, New York
  - Women'S Cancer Care Associates /ID# 269553, Albany, New York
  - Northwell Health Center for Advanced Medicine /ID# 269108, Lake Success, New York
  - NYU Laura and Isaac Perlmutter Cancer Center /ID# 269556, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 269529, New York, New York
  - University of North Carolina at Chapel Hill /ID# 269563, Chapel Hill, North Carolina
  - Duke Cancer Institute /ID# 269557, Durham, North Carolina
  - University of Cincinnati /ID# 269578, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center /ID# 269105, Columbus, Ohio
  - Kettering Medical Center /ID# 269585, Kettering, Ohio
  - Ou Health - Stephenson Cancer Center /ID# 269525, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute /ID# 269527, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute and Research Center /ID# 269988, Eugene, Oregon
  - Compass Oncology - Rose Quarter /ID# 270131, Portland, Oregon
  - Oregon Health and Science University /ID# 269581, Portland, Oregon
  - University Of Pittsburgh Medical Center Magee - Womens Hospital /ID# 269659, Pittsburgh, Pennsylvania
  - Allegheny Health Network West Penn Hospital /ID# 269551, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion /ID# 269574, Willow Grove, Pennsylvania
  - Sanford Cancer Center /ID# 269535, Sioux Falls, South Dakota
  - West Cancer Center and Research Institute - Germantown /ID# 269569, Germantown, Tennessee
  - Texas Oncology - Austin Central /ID# 269531, Austin, Texas
  - Texas Oncology - Bedford /ID# 269571, Bedford, Texas
  - Texas Oncology - Methodist Dallas Cancer Center /ID# 269554, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center /ID# 269532, Fort Worth, Texas
  - US Oncology Research Investigational Products Center /ID# 278746, Irving, Texas
  - Texas Oncology - San Antonio Medical Center - Research Drive /ID# 269549, San Antonio, Texas
  - University of Virginia Health System /ID# 269545, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk (Lake Wright) /ID# 269533, Norfolk, Virginia
  - VCU Health Adult Outpatient Pavillion /ID# 269570, Richmond, Virginia
  - Swedish Cancer Institute /ID# 269538, Seattle, Washington
- Argentina (4):
  - Sanatorio De La Mujer /ID# 269352, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires /ID# 269356, Buenos Aires
  - Hospital Italiano de Córdoba (Sociedad de Beneficencia Hospital Italiano) /ID# 269090, Córdoba
  - Isis Centro Especializado De Luce /ID# 269353, Santa Fe
- Australia (8):
  - Westmead Hospital /ID# 269362, Westmead, New South Wales
  - Gold Coast University Hospital /ID# 269365, Southport, Queensland
  - Ballarat Base Hospital /ID# 269364, Ballarat, Victoria
  - Monash Health - Monash Medical Centre /ID# 269360, Clayton, Victoria
  - Cabrini Hospital Malvern /ID# 269359, Malvern, Victoria
  - Peter MacCallum Cancer Centre /ID# 269361, Melbourne, Victoria
  - Epworth Hospital /ID# 269363, Richmond, Victoria
  - St. John Of God Subiaco Hospital /ID# 269358, Subiaco, Western Australia
- Belgium (7):
  - Imelda Ziekenhuis /ID# 269369, Bonheiden, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 269368, Brussels, Brussels Capital
  - Grand Hôpital De Charleroi - Notre Dame /ID# 269367, Charleroi, Hainaut
  - AZ Sint-Lucas /ID# 269366, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 269370, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 269091, Roeselare, West-Vlaanderen
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 269371, Namur
- Brazil (4):
  - Hospital Santa Izabel /ID# 269384, Salvador, Estado de Bahia
  - Catarina Pesquisa Clinica /ID# 269379, Itajaí, Santa Catarina
  - Beneficência Portuguesa de São Paulo /ID# 269092, São Paulo, São Paulo
  - Hospital Nove De Julho /ID# 269375, São Paulo, São Paulo
- Bulgaria (2):
  - Complex Oncology Center - Shumen /ID# 269372, Shumen
  - Comprehensive Cancer Center /ID# 269373, Vratsa
- Canada (12):
  - Arthur J. E. Child Comprehensive Cancer Centre /ID# 269388, Calgary, Alberta
  - Cross Cancer Institute /ID# 269392, Edmonton, Alberta
  - Bc Cancer Agency - Fraser Valley Centre /ID# 269398, Surrey, British Columbia
  - BC Cancer - Vancouver /ID# 269394, Vancouver, British Columbia
  - Juravinski Cancer Centre - Hamilton Health Sciences /ID# 269396, Hamilton, Ontario
  - Kingston General Hospital /ID# 269397, Kingston, Ontario
  - The Ottawa Hospital - General Campus /ID# 269391, Ottawa, Ontario
  - Princess Margaret Cancer Centre /ID# 269390, Toronto, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont /ID# 269395, Montreal, Quebec
  - CHUM - Centre hospitalier de l'Universite de Montréal /ID# 269387, Montreal, Quebec
  - McGill University Health Centre - Glen Site /ID# 269389, Montreal, Quebec
  - CIUSSS Estrie - Sherbrooke University Hospital Center /ID# 269393, Sherbrooke, Quebec
- China (26):
  - The first affiliated hospital of Bengbu medical college, Bengbu, Anhui
  - Capital Medical University (Cmu), Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University (Sysu) - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Province Cancer Hospital, Changsha, Hunan
  - The First Bethune Hospital Of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital Of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital Affliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital, Kunming, Yunnan
  - The Affiliated Women's Hospital Of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Czechia (4):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 269401, Brno, Brno-mesto
  - General University Hospital in Prague, Charles University /ID# 269402, Prague, Ceske Budejovice
  - Nemocnice Novy Jicin /ID# 269400, Nový Jičín, Novy Jicin
  - Fakultní nemocnice Ostrava /ID# 269403, Ostrava, Ostrava-mesto
- France (6):
  - Institut de cancérologie Strasbourg Europe (ICANS) /ID# 269419, Strasbourg, Bas-Rhin
  - Hôpital La Timone /ID# 269421, Marseille, Bouches-du-Rhone
  - Chu Dijon /Id# 269417, Dijon, Bourgogne-Franche-Comté
  - CHU Brest /ID# 269422, Brest, Finistere
  - Centre Leon Berard /ID# 269418, Lyon, Rhone
  - Institut Curie /ID# 269420, Paris, Île-de-France Region
- Germany (11):
  - Klinikum Esslingen /ID# 269435, Esslingen am Neckar, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg /ID# 269438, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 269439, Erlangen, Bavaria
  - Onkologische Schwerpunktpraxis Bielefeld /ID# 269440, Bielefeld, North Rhine-Westphalia
  - Universitaetsklinikum Bonn /ID# 269434, Bonn, North Rhine-Westphalia
  - Klinikum Dortmund Klinikzentrum Mitte /ID# 269441, Dortmund, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 269442, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 269433, Dresden, Saxony
  - Universitätsklinikum Gießen /ID# 269432, Giessen
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 269429, Hamburg
  - Krankenhaus Jerusalem /ID# 269430, Hamburg
- Greece (4):
  - St. Luke's Hospital S.A. /ID# 269445, Panórama, Thessaloniki
  - General Hospital of Athens Alexandra /ID# 269444, Athens
  - Hygeia Hospital /ID# 270132, Athens
  - IASO Hospital /ID# 269443, Marousi
- Ireland (7):
  - St James Hospital /ID# 269446, Dublin, Dublin
  - Bon Secours Cork Hospital /ID# 269449, Cork
  - Cork University Hospital /ID# 269451, Cork
  - Beaumont Hospital /ID# 269452, Dublin
  - University Hospital Galway /ID# 269447, Galway
  - Sligo General Hospital /ID# 269448, Sligo
  - Waterford Regional Hospital /ID# 269450, Waterford
- Israel (10):
  - Edith Wolfson Medical Center /ID# 269461, Holon, Central District
  - Meir Medical Center /ID# 269454, Kfar Saba, Central District
  - Rabin Medical Center /ID# 269456, Petah Tikva, Central District
  - Kaplan Medical Center /ID# 269457, Rehovot, Central District
  - The Chaim Sheba Medical Center /ID# 269094, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 269455, Tel Aviv, Tel Aviv
  - The Lady Davis Carmel Medical Center /ID# 269453, Haifa
  - Shaare Zedek Medical Center /ID# 269459, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 269458, Jerusalem
  - ZIV Medical Center /ID# 269460, Safed
- Italy (21):
  - Azienda Ospedaliero Universitaria Careggi /ID# 269465, Florence, Firenze
  - Ente Ospedaliero Ospedali Galliera /ID# 269472, Genoa, Genova
  - Ospedale San Martino /ID# 269469, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 269473, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 269475, Milan, Milano
  - Istituto Nazionale Dei Tumori /ID# 269477, Milan, Milano
  - Casa di Cura San Pio X /ID# 277973, Milan, Milano
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale /ID# 269097, Naples, Napoli
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 269474, Meldola, Reggio Emilia
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 269470, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 269096, Rome, Roma
  - Ospedale di Mirano - Azienda ULSS 3 /ID# 269462, Mirano, Venezia
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 269476, Bologna
  - Ospedale Cannizzaro /ID# 269478, Catania
  - Alessandro Manzoni Hospital /ID# 269467, Lecco
  - Azienda USL Toscana Nord Ovest - Ospedale San Luca /ID# 269095, Lucca
  - Azienda Ospedaliero Universitaria Di Parma /ID# 269466, Parma
  - Fondazione IRCCS Policlinico San Matteo /ID# 269463, Pavia
  - AUSL Piacenza-Ospedale Guglielmo da Saliceto /ID# 269468, Piacenza
  - New Hospital of Prato - S. Stefano /ID# 269464, Prato
  - AUSL di Reggio Emilia - Arcispedale Santa Maria Nuova /ID# 269471, Reggio Emilia
- Japan (22):
  - Aichi Cancer Center /ID# 274332, Nagoya, Aichi-ken
  - Chiba University Hospital /ID# 274371, Chiba, Chiba
  - The Jikei University Kashiwa Hospital /ID# 274334, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center /ID# 276078, Matsuyama, Ehime
  - Kurume University Hospital /ID# 274337, Kurume-shi, Fukuoka
  - Sapporo Medical University Hospital /ID# 274330, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 274331, Sapporo, Hokkaido
  - Hyogo Cancer Center /ID# 274323, Akashi-shi, Hyōgo
  - Iwate Medical University Hospital - Yahabacho /ID# 274635, Yahaba, Iwate
  - Kagoshima University Hospital /ID# 276081, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 274336, Isehara, Kanagawa
  - Tohoku University Hospital /ID# 274327, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 274329, Niigata, Niigata
  - Okayama University Hospital /ID# 274324, Okayama, Okayama-ken
  - Osaka Medical And Pharmaceutical University Hospital /ID# 276079, Takatsuki, Osaka
  - Saitama Medical University International Medical Center /ID# 274953, Hidaka, Saitama
  - Shizuoka Cancer Center /ID# 274325, Sunto-gun, Shizuoka
  - Jichi Medical University Hospital /ID# 274634, Shimotsuke-shi, Tochigi
  - National Cancer Center Hospital /ID# 274321, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 274326, Koto-ku, Tokyo
  - Keio University Hospital /ID# 276159, Shinjuku-ku, Tokyo
  - The Jikei University School of Medicine /ID# 276160, Tokyo
- Philippines (3):
  - The Medical City /ID# 269493, Pasig, National Capital Region
  - East Avenue Medical Center /ID# 269099, Quezon City, National Capital Region
  - Cardinal Santos Medical Center /ID# 269100, San Juan City, National Capital Region
- Poland (4):
  - Wielkopolskie Centrum Onkologii /ID# 269494, Poznan, Greater Poland Voivodeship
  - Jagiellonskie Centrum Innowacji Sp. z o.o. /ID# 269497, Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewodzki im. Sw. Jana Pawla II w Siedlcach Sp. z o.o. /ID# 269500, Siedlce, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o.o. /ID# 269495, Gdynia, Pomeranian Voivodeship
- South Korea (12):
  - National Cancer Center /ID# 269481, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 269489, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 269482, Seongnam-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 269488, Daegu, Gyeongsangbuk-do
  - Korea University Anam Hospital /ID# 269486, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 269479, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 269483, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 269480, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 269484, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 269487, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 269485, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 269490, Seoul, Seoul Teugbyeolsi
- Spain (11):
  - Complejo Hospitalario Universitario A Coruña /ID# 269414, A Coruña, A Coruna
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 269409, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia /ID# 270296, Córdoba, Cordoba
  - Hospital Universitario Virgen de la Victoria /ID# 269413, Málaga, Malaga
  - Clinica Universidad de Navarra - Pamplona /ID# 269410, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron /ID# 269406, Barcelona
  - Hospital Clinic de Barcelona /ID# 269408, Barcelona
  - Hospital Universitari De Girona Doctor Josep Trueta /ID# 269411, Girona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 269405, Madrid
  - Hospital Universitario La Paz /ID# 269407, Madrid
  - Hospital Clínico Universitario de Valencia /ID# 269412, Valencia
- Turkey (Türkiye) (3):
  - Baskent Universitesi Adana Uyg. Ve Arast. Merkezi Yuregir Baskent Hastanesi /ID# 270174, Adana
  - Hacettepe University Faculty of Medicine /ID# 269521, Ankara
  - Başkent Üniversitesi Ankara Hastanesi /ID# 269524, Ankara
- United Kingdom (8):
  - Cheltenham General Hospital /ID# 269427, Cheltenham, Gloucestershire
  - Guy's Hospital /ID# 269426, London, Greater London
  - The Royal Marsden - Chelsea /ID# 269102, London, Greater London
  - Mount Vernon Hospital /ID# 269423, Northwood, Greater London
  - University Hospital Southampton /ID# 269425, Southampton, Hampshire
  - The Royal Marsden - Sutton /ID# 269103, Sutton, Surrey
  - The Christie /ID# 269428, Manchester
  - Singleton Hospital /ID# 269424, Swansea

REFERENCES:
- [Derived] O'Malley DM, Myers T, Wimberger P, Van Gorp T, Redondo A, Cibula D, Nicum S, Rodrigues M, Backes FJ, Barlin JN, Lewin SN, Lim P, Pothuri B, Diver E, Banerjee S, Lorusso D. Maintenance with mirvetuximab soravtansine plus bevacizumab vs bevacizumab in FRalpha-high platinum-sensitive ovarian cancer. Future Oncol. 2024;20(32):2423-2436. doi: 10.1080/14796694.2024.2372241. Epub 2024 Jul 31. PMID 39082675
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN853-0421